CLINICAL TRIAL: NCT04667182
Title: Meal-centric Insulin Dosing for Optimized Post-Prandial Glucose Control in People Using Multiple Daily Injections
Brief Title: A Study of Glucose Control in Participants With Type 1 and Type 2 Diabetes
Status: Withdrawn | Type: Observational
Why Stopped: Study was withdrawn prior to enrolment due to business decision.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 17420; F3Z-MC-IORN (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-12-11; First posted 2020-12-14 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
Keywords: T1D; T2D
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Fitness Trackers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Combined Diabetes Management Data: Participants with type 1 and type 2 diabetes will use a meal tagging application (app) and fitness tracker. They will upload these data to a web portal where they will be matched with data from their insulin pen and continuous glucose monitor (CGM). Combined data will be used as a complement to standard of care for diabetes management.
  Interventions: Other: Meal-Tagging App and Web-based Portal:; Device: Fitness Tracker

INTERVENTIONS:
Other: Meal-Tagging App and Web-based Portal: — Meal tagging app to capture frequently eaten meals and test meals for 18 weeks.
Device: Fitness Tracker — Fitness tracker will be worn around the clock for 18 weeks.

SUMMARY:
The main purpose of this study is to determine whether combining meal, glucose and insulin data in a web-based system will improve management of type 1 (T1D) and type 2 diabetes (T2D). No study drug will be given. The study will last about 18 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with type 1 or type 2 diabetes for >3 years by clinical diagnosis who use basal insulin, in addition to at least one injection of meal time insulin per day
* Insulin pen use for at least 3 months
* Current use of or willingness to use Dexcom G6 at least 6 out of 7 days per week
* A1c 6.5-9.5%

Exclusion Criteria:

* Currently using any form of insulin pump, including hybrid closed-loop system (e.g., Medtronic 670G)
* Individuals requiring single insulin boluses of >40 units
* Individuals planning to follow a specific diet plan for weight loss
* Inability to consume regular, consistent meals
* Individuals who have had severe hypoglycemia with seizure or coma within the past 6 months
* Individuals who have been hospitalized for diabetic ketoacidosis (DKA) within the past 6 months

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with T1D and T2D
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-01-25 (Estimated); Primary Completion 2021-12-06 (Estimated); Study Completion 2021-12-06 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Area Under the Curve (AUC) of CGM | Baseline, Week 17
  Change from Baseline in AUC of CGM

SECONDARY OUTCOMES:
Qualitative data from study investigators and participants | Baseline through Week 17
  Qualitative data describing experience from study investigators and participants
Percent Time-in-Range (TIR) | Baseline through Week 17
  Percent Time-in-Range defined as glucose >70 and ≤180 milligrams per deciliter [mg/dL])
Postprandial TIR | Baseline through Week 17
  Postprandial TIR is defined as TIR glucose: glucose >=70 and ≤180 mg/dL
Time Above Range (TAR) | Baseline through Week 17
  TAR is defined as glucose > 180 mg/dL
Time Below Range (TBR) <70 mg/dL | Baseline through Week 17
  TBR is defined as glucose < 70 mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (2):
- United States (2):
  - Boston Medical Center, Boston, Massachusetts
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No